CLINICAL TRIAL: NCT04017091
Title: The Impact of Virtual Reality Training on Executive and Complex Attentional Functions and Association With Neurorehabilitation Outcomes
Brief Title: Neurocognitive Rehabilitation Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 014-083
Record Dates: First submitted 2019-06-19; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Acquired Brain Injury
Keywords: Virtual Reality Exposure Therapy; Executive Function; Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Mixed design study with quasi-experimental Intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VR Group (Experimental): ABI Patients Twenty-one patients with ABI participated in this pilot study (Figure 1): 9 diagnosed with stroke (43%), 6 with TBI (29%), 2 with anoxic injury (10%), 3 with brain tumor (14%), and 1 with amyloid angiopathy (5%).
  Interventions: Diagnostic Test: Virtual Reality Cognitive Training
- Control Group (Standard Care) (No Intervention): The 12 Controls were age- and gender-matched (and etiology when possible) patients who had previously received traditional neurorehabilitation and completed the same measures as the VR group prior to onset of the study, but they did not receive VR treatment.

INTERVENTIONS:
Diagnostic Test: Virtual Reality Cognitive Training — Bimodal VR-Stroop (ClinicaVR: Apartment Stroop) Patient find themselves seated with a virtual apartment, where they see a living room, in front of a flat-screen TV set, a kitchen and a window. This intervention consisted of two Stroop conditions across all 8 sessions. In Condition 1 (Inhibition), Patients indicated when the color named (audio stimulus) matched the color shown (visual stimulus). Participants were to withhold their response in mismatched trials. In Condition 2 (Interference), Participants clicked the mouse when the color heard was the same as the ink color; not the word printed.
  Other Names: VR Group
  Arms: VR Group

SUMMARY:
Objective: To determine whether immersive virtual reality (VR) treatment interventions improve executive dysfunction and complex attention deficits in patients with brain injury compared with standard neurorehabilitation, and whether VR performance predicts neurorehabilitation outcomes at discharge.

Design: Mixed design study with quasi-experimental Intervention group (N = 12) and retrospective Control group (N = 12). Both groups were compromised of individuals with brain injury admitted to an outpatient day neurorehabilitation program.

DETAILED DESCRIPTION:
The current study focuses on repeated practice of a VR-based cognitive intervention with the intent of improving cognitive deficits known to impact ability to resume complex activities. This study details implementation of VR within a neurorehabilitation setting. Associations between the VR Stroop and neuropsychological, speech therapy, and global rehabilitation measures are examined. The investigators include a brain injured control group to address this frequently cited methodological concern.

Inclusion Criteria Patients participating in this study were aged 18 years and older diagnosed with acquired traumatic or non-traumatic neurologic illness, and with dysfunction in executive and attention skills documented during their inpatient rehabilitation course.

Patients that had not yet undergone a neuropsychological evaluation by the time they consented to participate in the study, were administered the Orientation and Cognitive Log (OLOG/Cog-Log) to ensure they were oriented and had sufficient cognitive ability to attend to and understand instructions.

Exclusion Criteria Patients were excluded from participating in the study if they were medically unstable, as deemed by their primary doctor, were aphasic or had hemispatial neglect, had prior history of significant neurological complications or developmental delay resulting in compromised cognition, prisoners, and if they did not speak English.

Participants ABI Patients Twenty-one patients with ABI participated in this pilot study (Figure 1): 9 diagnosed with stroke (43%), 6 with TBI (29%), 2 with anoxic injury (10%), 3 with brain tumor (14%), and 1 with amyloid angiopathy (5%). Six of the 21 patients partially completed the study, but failed to complete all 8 intervention sessions. Two patients were medically withdrawn from Day Neuro due to refractory medical complications, two patients self-discharged from the program against medical advice, and two patients' rehabilitation regimens were concluded prior to their projected discharge dates when insurance or state-assisted benefits were not extended. Of the remaining 15 participants, 12 completed neuropsychological evaluation. The final analyses included 12 patients with ABI who completed VR treatment and all neuropsychological and rehabilitation outcome measures, and 12 Controls with ABI (see Figure 1).

Control Group The 12 Controls were age- and gender-matched (and etiology when possible) patients who had previously received traditional neurorehabilitation and completed the same measures as the VR group prior to onset of the study, but they did not receive VR treatment. Their data was obtained via retrospective chart review of patients admitted to Day Neuro between 04/2013 and 07/2014.

Intervention Schedule Patients completed the VR apartment program twice per week for a 4-week period (8 sessions total). The VR interventions replaced 30-60 minutes of speech therapy and/or 30-60 minutes of independent time (time designated for relaxation or completion of therapy assignments) per week of the study. Otherwise, clinical services were not altered (see Appendix 1 for detailed schedule of VR and Day Neuro therapy regimen).

The total duration of sessions 1 and 8 was approximately 60 minutes each. The duration of sessions 2-7 was 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Diagnosis of acquired traumatic or non-traumatic neurologic illness
* Documented dysfunction in executive and attention skills
* OLOG/Cog-Log score ≥ 25/30

Exclusion Criteria:

* Medically unstable (as deemed by primary doctor)
* Aphasic
* Hemispatial neglect
* Prior history of significant neurological complications
* Prior history of developmental delay resulting in compromised cognition
* Prisoners
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
VR Stroop: Change in response times from session1 to session 8 for correct and incongruent trials | 2 times a week for 4 weeks. VR Stroop is administered during all sessions: sessions 1-8
  The VR Stroop was administered at each of the 8 study sessions, through study completion. In both the Inhibition and the Interference Trial, the metric being measured was how quickly patient responds to a target on matching (visual color matches aurally presented color) and non-matching trials (visual color does not match aurally presented color). Metric is measured in milliseconds.
VR Stroop: Change in number of total commission errors | 2 times a week for 4 weeks. VR Stroop is administered during all sessions: sessions 1-8
  The VR Stroop was administered at each of the 8 study sessions, through study completion. In both the Inhibition and the Interference Trial, the metric being measured was # of impulsive responses (raw score).
VR Stroop: Change in number of total omission errors | 2 times a week for 4 weeks. VR Stroop is administered during all sessions: sessions 1-8
  The VR Stroop was administered at each of the 8 study sessions, through study completion. In both the Inhibition and the Interference Trial, the metric being measured was # of attentional errors (missed items raw score).

SECONDARY OUTCOMES:
Wechsler Test of Adult Reading (WTAR) | After week 4 of study - which was typically week 5-7 of the neurorehabilitation course (Administration of traditional neuropsychological measures followed study completion to avoid confounds & practice effects). Single time point.
  The WTAR is a single-word reading or word pronunciation measure. It also provides an estimate of premorbid intellectual functioning. The metric of interest for the WTAR was the total score (standard score). In statistics, the standard score is the signed number of standard deviations an observation or datum is above the mean. The mean standard score for the WTAR is 100, with scores above the mean being positive, and scores below the mean being negative. This data was archival for Controls.
Trail Making Tests (TMT) | After week 4 of study - which was typically week 5-7 of the neurorehabilitation course (Administration of traditional neuropsychological measures followed study completion to avoid confounds & practice effects). Single time point.
  TMT measures visuomotor processing speed, visual attention, and set-shifting. The raw score was time to completion in seconds, with lower values indicating stronger performance and higher values indicating weaker performance. This raw score was converted to a T-score. We also analyzed number of raw errors (reversals and set-shifting). This data was archival for Controls.
Verbal Fluency Tests (COWAT and Animals) | After week 4 of study - which was typically week 5-7 of the neurorehabilitation course (Administration of traditional neuropsychological measures followed study completion to avoid confounds & practice effects). Single time point.
  COWAT assess phonemic fluency. Animals assessed category fluency. The raw score consists of total number correct across 3 trials for COWAT and a single trial for Animals. The raw score is converted to a T-score. This data was archival for Controls.
Stroop Color and Word Test, Golden version | After week 4 of study - which was typically week 5-7 of the neurorehabilitation course (Administration of traditional neuropsychological measures followed study completion to avoid confounds & practice effects). Single time point.
  The Golden version Stroop consists of 3 trials: word reading, color naming, and inhibition. The raw score consists of the number of words or colors correctly read within 45 seconds. Lower values indicate stronger performance and higher values indicate weaker performance. The raw score for each trial is converted to a T-score. This data was archival for Controls.
Functional Assessment of Verbal Reasoning and Executive Strategies (FAVRES) | Week 1 of study and after week 4 of study.
  Performance on the Make a Decision subtest: Accuracy Raw and Analysis of Reasoning Raw scores. Accuracy of the solution to each sub-test is scored on a scale from 0 (no viable solution) to 5 (best possible solution). Reasoning (rationale) is based on # of valid reasons included in response, with raw score equaling the # of viable options. This data was archival for Controls.
Ross Information Processing Assessment (RIPA), 2nd Edition | Week 1 of study and after week 4 of study.
  Problem-Solving subtest raw score: Patient is required to respond to 10 stimuli requiring problem-solving and reasoning strategies for task completion. Organization subtest raw score: Patient is required to recall category members within a 1-minute time limit and to recall a category type given three category members. More response options generated indicates stronger performance for both subtests, with a raw score out of a maximum of 30 (X/30). This data was archival for Controls.
Holistic Outcome Measure (HOM): Change in level of independence | HOM home, community, and community participation scores at discharge compared with those at admission.
  The HOM assess level of independence in (1) the home, (2) the community, and (3) community participation, rated 1-5 by clinicians. A score of 1 indicates a need for full-time supervision and participation is limited to medical appointments, and 5 indicates full independence. Each category is considered independently. This data was archival for Controls.
Mayo-Portland Adaptability Inventory, 4th Edition (MPAI-4): Change in level of independence | MPAI-4 abilities, adjustment, and participation scores at discharge compared with those at admission.
  MPAI-4 consists of 3 subscales: Abilities, Adjustment, Participation, which assess sensory, cognitive, and motor abilities; emotional and neurological symptoms, interpersonal adjustment, and awareness; & social, work, and leisure participation and management of IADLs respectively. They are rated 0-4 by clinician (0 = No problem, does not interfere with activities; does not use assistive device or medication; 4 = Severe problem; interferes with activities more than 75% of the time). Each subscale is summed to produce a score, and all 3 subscores are combined to produce a total score. This data was archival for Controls.

OTHER OUTCOMES:
Simulator Sickness Questionnaire (SSQ) | 6 time intervals over 4 weeks (1x in week 1, 2x in week 2, 2x in week 3, 1x in week 4). During VR sessions 2-7.
  The SSQ assesses occurrence, nature and severity of sickness symptoms induced by VR environment, rated 0-3 by patient. A score of indicates =no symptom; 1=slight; 2=moderate; 3=severe symptoms. As such, lower scores indicate that a patient is less affected by the use of VR devices.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Dahdah, Ph.D., Principal Investigator — Baylor Scott and White Institution for Rehabilitation

IPD SHARING:
Plan to Share IPD: No